CLINICAL TRIAL: NCT05970523
Title: Investigation of the Effects of Core Stabilization Exercises on Balance, Trunk Muscle Endurance and Posture in Healthy Sedentary Individuals
Brief Title: The Effects of Core Stabilization Exercises on Balance, Trunk Muscle Endurance and Posture on Sedentary Individuals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Beyza Nur Yumak, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-772.02-2555
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Core Stabilization; Sedentary Behavior
Keywords: Trunk Muscle Endurance; Balance; Posture
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: I applied exercise intervention for the intervention group. I will not apply any intervention for the control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Intervention includes core stabilization exercises for 45 minutes 3 times a week. Participants do exercise face to face under supervision of a physiotherapist and via an online application under the supervision of a physiotherapist once a week. Also participants do home exercise once a week. Exercise group walk for an hour in other two days.
  Interventions: Other: Core Stabilization Exercises
- Control Group (No Intervention): There is no exercise or intervention for control group.

INTERVENTIONS:
Other: Core Stabilization Exercises — Core stabilization exercises are known as a very effective exercise method based on the motor learning principle, performed with the individual's own body weight to strengthen the muscles, improve balance, posture, trunk muscle endurance and flexibility.Each exercise was performed for 7-8 seconds with 10 repetitions. Progression in the exercises was achieved by increasing the difficulty level of the exercises according to the participant's condition once every two weeks.
  Arms: Exercise Group

SUMMARY:
There are very few studies on the effect of core stabilization exercises on balance, posture and trunk muscle endurance in healthy sedentary individuals in literature. The goal of the study is to investigate the effects of core stabilization exercises on balance, trunk muscle endurance and posture in healthy sedentary individuals. According to the results of International Physical Activity Questionnaire, the researcher includes sedentary individuals over the age of 18 in the study. The participants are divided into two groups as control (n=21) and exercise (n=21) groups. The outcome measures are The Stabilizer Pressure Biofeedback Unit, New York Posture Assesment Scale, Korebalance Balance System, trunk muscle endurance tests. Intervention includes core stabilization exercises 3 times a week and walking twice a week for 6 weeks. There is no treatment or intervention for the control group. The researcher evaluates both groups at the beginning and 6 weeks after the intervention.

DETAILED DESCRIPTION:
Core stabilization exercises are performed under the supervision of a physiotherapist as face-to-face exercises, guided online exercises, and as an individual home exercise each once a week, totaling 3 times a week. Each exercise will be performed with 10 repetitions for 8 seconds. Each of the exercises is varied from easy to difficult. Progress in the exercises will be achieved by increasing the difficulty level of the exercises according to the condition of the participant once every two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be voluntary to participate in the study
* Being between the ages of 18-40
* Being sedentary

Exclusion Criteria:

* Not volunteering to participate in the study
* Having a complaint of low back pain in the last two months
* Being pregnant
* Having chronic lower extremity pain
* Having an orthopedic disease and undergoing a surgical operation
* Having had abdominal surgery
* Being a neurological disease pathology

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
New York Posture Assessment Scale | 6 weeks
  This test assesses alignment of various body parts of an individual in anatomical position. The New York Posture Rating Scale detects postural changes. There are 3 figure drawings for each of the 13 different body parts that provide general postural alignment. In the evaluation, five (5) points are given if the person's posture is correct, three (3) points if moderately impaired, and one (1) point if severely impaired. At the end of the evaluation, the total maximum score is 65 and the minimum is 13. Postural disturbances increase as the score decreases.
KoreBalance Balance System | 6 weeks
  The Korebalance Balance System is a computerized balance and exercise system. The software of the system assigns a score following static and dynamic balance evaluations. As stated in the device manual, a score of 700 and below was considered normal and above was considered risky for static balance and a score of 2000 and below was considered normal and above was considered risky for dynamic tests. A higher score is associated with more balance disorders.
Trunk Muscle Endurance Tests | 6 weeks
  The endurance of the trunk flexor, trunk extensor and lateral flexor muscles is evaluated by recording the maximum time that the person can maintain the test position. Measurements are made using a stopwatch and the result is recorded in seconds. The tests are repeated twice to save the best measurement value. Tests are terminated when the participant's position deteriorates or when the participant says cannot continue the test.
International Physical Activity Questionnaire | Before Intervention (First Assesment)
  This survey lists activities and requests estimates of duration and frequency for each activity performed in the past week. The times are multiplied by the known Metabolic Equivalents (METs) per activity and the results for all items are summed, resulting in the overall physical activity score.

SECONDARY OUTCOMES:
The Stabilizer Pressure Biofeedback Unite | 6 weeks
  This device evaluates contraction of deep abdominal muscles, muscle activity and segmental stability. The device has values between 0 mmHg and 200 mmHg, varying in intervals of 2 mmHg. Movement or change in position causes volume changes in the pressure bag.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Nur Tunali, Professor, Study Director — Medipol University
Locations (1):
- Beyza Nur Yumak, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sekendiz B, Cug M, Korkusuz F. Effects of Swiss-ball core strength training on strength, endurance, flexibility, and balance in sedentary women. J Strength Cond Res. 2010 Nov;24(11):3032-40. doi: 10.1519/JSC.0b013e3181d82e70. PMID 20940644
- [Result] Hung KC, Chung HW, Yu CC, Lai HC, Sun FH. Effects of 8-week core training on core endurance and running economy. PLoS One. 2019 Mar 8;14(3):e0213158. doi: 10.1371/journal.pone.0213158. eCollection 2019. PMID 30849105
- [Result] von Garnier K, Koveker K, Rackwitz B, Kober U, Wilke S, Ewert T, Stucki G. Reliability of a test measuring transversus abdominis muscle recruitment with a pressure biofeedback unit. Physiotherapy. 2009 Mar;95(1):8-14. doi: 10.1016/j.physio.2008.10.003. Epub 2009 Jan 22. PMID 19627680
- [Result] Dogruoz Karatekin B, Yasin S, Yumusakhuylu Y, Bayram F, Icagasioglu A. Validity of the Korebalance(R) Balance System in Patients with Postmenopausal Osteoporosis. Medeni Med J. 2020;35(2):79-84. doi: 10.5222/MMJ.2020.18828. Epub 2020 Jun 30. PMID 32733755
- [Result] Evans K, Refshauge KM, Adams R. Trunk muscle endurance tests: reliability, and gender differences in athletes. J Sci Med Sport. 2007 Dec;10(6):447-55. doi: 10.1016/j.jsams.2006.09.003. Epub 2006 Dec 1. PMID 17141568
- [Result] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606